CLINICAL TRIAL: NCT02728388
Title: Topical Photodynamic Therapy (PDT) With Levulan® Kerastick® for Benign Dermal Neurofibromas Phase II
Brief Title: Photodynamic Therapy for Benign Dermal Neurofibromas- Phase II
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Donald Basel (Other)
Responsible Party: Sponsor-Investigator, Donald Basel, Professor, Medical College of Wisconsin
Organization: Medical College of Wisconsin (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00026795
Record Dates: First submitted 2016-03-25; First posted 2016-04-05 (Estimated); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: NEUROFIBROMATOSIS 1
Keywords: NF1; Neurofibroma; Neurofibromatosis Type 1
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma | interventions — Aminolevulinic Acid; Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PDT Treatment (Experimental): Each subject will have either placebo or Levulan Kerastick topical application applied to matched sets of neurofibromas. Each subject will have both sets, in order to serve as his/her own control subject.
  16 to 24 hours post study drug treatment, both sets of neurofibromas, Levulan and placebo treated, will be irradiated with red light (630 nm) from an Omnilux Revive light device at 100 mW/cm2 for 1000 seconds (16.7 minutes).
  Interventions: Drug: aminolevulinic acid

INTERVENTIONS:
Drug: aminolevulinic acid — Drug: Levulan Kerastick
  Drug: Topical placebo
  Device: Omnilux Revive
  Procedure: Photodynamic therapy
  Other: Tumor growth rate measurements
  Other Names: Photodynamic therapy

SUMMARY:
The investigators wish to determine the time to disease progression for benign neurofibromas treated with Levulan Kerastick topical photosensitizer and red light photodynamic therapy (PDT) in patients with neurofibromatosis type 1 (NF1).

The investigators also wish to measure tumor size for control and treatment tumors in order to gain insights into tumor growth rates.

DETAILED DESCRIPTION:
Neurofibromas contain a large quantity of fibrous matter, and it is not anticipated that significant reductions in tumor size can be achieved in large, long established, tumors. Cutaneous neurofibromas, which do not usually become apparent until puberty, continue to increase in size and number throughout adulthood. The psychosocial burden of these disfiguring tumors is significant, and the targeted age group (14-30) is at a life period associated with an acceleration in tumor growth. It is for these reasons that the investigators hope to affect the growth rate of less established tumors, in order to prevent or lessen this burden as the patient progresses further into adulthood.

Therefore, the investigators wish to determine the time to disease progression (defined as 50% growth in size over baseline) for benign neurofibromas treated with PDT in patients with neurofibromatosis type 1 (NF1) in subjects aged 14-30.

The treatment will consist of choosing several neurofibromas of similar size, and applying a topical drug called Levulan, or just the topical application alone (a placebo). Within 24 hours of drug treatment, the neurofibromas will be illuminated with red light (both Levulan and placebo). The Levulan is what is known as a photosensitizer, and will be activated by the red light to potentially kill some of the tumor cells. Approximately every 6 months after, for three years, the tumors will be measured by digital photography and ultrasound to see if they are growing more slowly than the ones with the placebo application alone.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 14 years or older.
2. Diagnosed NF1, determined by American Academy of Neurology Guidelines (see Diagnosis section).
3. Tumor Location: cutaneous, trunk, or limbs only.
4. Tumor Type: superficial dermal neurofibromas ≤4mm deep.
5. Patient has provided written informed consent.
6. Patient is willing to and can comply with study follow-up requirements.
7. Absence of any other malignancy.

Exclusion Criteria:

1. Life expectancy less than 3 years.
2. Pregnancy.
3. Cutaneous photosensitivity to the wavelengths used to active PDT.
4. A diagnosis of porphyria.
5. Allergy to aminolevulinic acid or any of the topical solution vehicle components.
6. Previous chemotherapy within 6 weeks of proposed PDT.
7. Other concurrent tumor therapy.

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Time to disease progression | 3 years
  The time it takes for 50% growth in tumor size over baseline measurements.

SECONDARY OUTCOMES:
Tumor growth rate | 3 years
  Measure tumor size for control and treatment tumors in order to gain insights into tumor growth rates.

CONTACTS AND LOCATIONS:
Overall Officials: Donald G Basel, MD, Study Director — Medical College of Wisconsin
Locations (1):
- Donald G Basel, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No